CLINICAL TRIAL: NCT00014599
Title: Phase II Clinical Trial On Taxol As Single Agent In Locally Advanced And/Or Metastatic Or Recurrent Vulva Cancer Not Amenable For Surgery And/Or Radiotherapy
Brief Title: Paclitaxel in Treating Patients With Locally Advanced, Metastatic, or Recurrent Cancer of the Vulva
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-55985; EORTC-55985
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Vulvar Cancer
Keywords: stage III vulvar cancer; stage IV vulvar cancer; recurrent vulvar cancer; squamous cell carcinoma of the vulva
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients who have locally advanced, metastatic, or recurrent cancer of the vulva.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic activity of paclitaxel in patients with locally advanced, metastatic, or recurrent squamous cell carcinoma of the vulva.
* Determine the objective response rate and duration of response in these patients treated with this drug.
* Determine the acute side effects of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 21 days for a maximum of 10 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 9 weeks.

PROJECTED ACCRUAL: A total of 16-29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the vulva

  * Not suitable for radiotherapy or surgery as first-line treatment
* Measurable or evaluable disease

  * At least 1 bidimensionally measurable target lesion
  * Measurable metastatic disease outside previously irradiated areas OR
  * Local recurrence within a previously treated area OR
  * Local lesions showing progression while on treatment
* No brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2
* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT less than 2 times upper limit of normal

Renal:

* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No prior or concurrent cardiac disease (i.e., uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the past year, cardiac ventricular arrhythmia requiring medication, or 2nd or 3rd degree heart block)

Other:

* No peripheral neuropathy greater than grade 1
* No serious active infection
* No prior allergic reaction to drugs containing Cremophor EL
* No other serious medical, psychological, familial, or social condition that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy except as concurrent therapy with radiotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* See Chemotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-02; Primary Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Els Witteveen, MD, PhD, Study Chair — UMC Utrecht
Locations (14):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Centre Henri Becquerel, Rouen, France
- Italy (4):
  - European Institute of Oncology, Milan
  - Ospedale Mauriziano Umberto I, Torino
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Civile, Voghera
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - University Medical Center Nijmegen, Nijmegen
  - Academisch Ziekenhuis Utrecht, Utrecht
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- United Kingdom (3):
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Oldchurch Hospital, Romford, England
  - Western Infirmary, Glasgow, Scotland

REFERENCES:
- [Result] Witteveen PO, van der Velden J, Vergote I, Guerra C, Scarabeli C, Coens C, Demonty G, Reed N. Phase II study on paclitaxel in patients with recurrent, metastatic or locally advanced vulvar cancer not amenable to surgery or radiotherapy: a study of the EORTC-GCG (European Organisation for Research and Treatment of Cancer--Gynaecological Cancer Group). Ann Oncol. 2009 Sep;20(9):1511-1516. doi: 10.1093/annonc/mdp043. Epub 2009 Jun 1. PMID 19487487